CLINICAL TRIAL: NCT04332601
Title: Assessment of the Efficacy of a Fatigue Management Therapy in Schizophrenia: a Randomized Controlled Multi-centric Study
Brief Title: Assessment of the Efficacy of a Fatigue Management Therapy in Schizophrenia
Acronym: ENERGY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7778
Record Dates: First submitted 2020-03-11; First posted 2020-04-02 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia
Keywords: fatigue; schizophrenia; microbiota; cognitive behavioral therapy
MeSH Terms: conditions — Schizophrenia; Fatigue | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENERGY intervention (Experimental): ENERGY Intervention:
  * 14 sessions of 1h CBT intervention (standardized fatigue treatment comprising six modules over 14 individual therapy sessions)
  * 1 session per week
  * With a psychologist (different to the psychologist who will perform the assessments)
  * Individual sessions
  * and Treatment as usual
  Interventions: Behavioral: Fatigue Management Therapy
- Treatment as usual (TAU) (Other): * Comparison group
  * TAU defined by antipsychotic medication coupled with day hospital care
  Interventions: Other: TAU (Treatment as usual)

INTERVENTIONS:
Behavioral: Fatigue Management Therapy — 14 sessions of 1h CBT intervention
  Arms: ENERGY intervention
Other: TAU (Treatment as usual) — No CBT intervention
  Arms: Treatment as usual (TAU)

SUMMARY:
Fatigue is commonly experienced in numerous pathologies, including schizophrenia. Research has shown that chronic fatigue can exacerbate clinical symptoms.

Several evidence-based interventions for fatigue syndrome have been shown to be effective in other medical conditions, but up to this date no research has assessed interventions in fatigue management within psychotic populations.

The aim of this study is to evaluate (in a multisite single blind randomized clinical trial) the efficacy of a cognitive-behavioral therapy (CBT) intervention of fatigue management in people diagnosed with schizophrenia. Secondary objectives include the examination of changes in fatigue scores as well as clinical symptoms, physical & cognitive functioning, quality of life at 9-month post CBT intervention. Another aim in this study is to assess - MICROBIATE

The investigators hypothesize that following the CBT treatment intervention, patients will demonstrate reduced level of fatigue. No change in the severity of fatigue is expected in the group receiving treatment as usual.

ELIGIBILITY:
Inclusion criteria:

1. Aged between 18 and 60 years,
2. patients with a diagnosis of schizophrenia according to DSM 5 validated after a clinical evaluation by one psychiatrist investigators,
3. patients with a score at the 4th subscale of "Multidimensional Fatigue Inventory " greater or equal to 10
4. patients with a follow-up in a day hospital at inclusion,
5. subjects must be able to attend all scheduled visits and comply with all trial procedures,

Non inclusion criteria:

1. subject unable to read or/and write French,
2. planned long-term stay outside of the study region that prevents compliance with the visit plan,
3. patients with a history of severe brain trauma,
4. patients with a history of neurological pathology,
5. patients pregnant or breast-feeding
6. patients deprived of liberty
7. patients participating in another ongoing biomedical study
8. patients not affiliated with a French social security scheme or beneficiary of such a scheme
9. Absence of signed informed consent form by the patient and the patient's tutor if he has one

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory (MFI) | Change between baseline and 3 months later (corresponding to the end of the treatment intervention)
  MFI - self-assessment instrument with 20 items including 5 dimensions: General, Physical, and Mental Fatigue, Reduced Motivation and Reduced Activity

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | baseline - 3 months - 9 months
  PANSS - 30 item scale assessing level of symptomatology (positive, negative, general psychopathology) in psychotic disorders
Clinical Assessment Interview for Negative Symptoms (CAINS) | baseline - 3 months - 9 months
  CAINS - semi-structured interview measuring level of severity of negative symptoms
Calgary Depression Scale for Schizophrenia (CDSS) | baseline - 3 months - 9 months
  CDSS - 9 item scale assessing level of depressive symptomatology in schizophrenic populations
Berlin Questionnaire (BQ) | baseline - 3 months - 9 months
  BQ- questionnaire consisting of 3 categories related to the risk of having sleep apnea; snoring (section 1), daytime somnolence (section 2), and hypertension and BMI (section 3
Idiopathic Hypersomnia Severity Scale (IHSS) | baseline - 3 months - 9 months
  IHSS - self-report measure of 14 items assessing - hypersomnolence symptoms, consequences, and responsiveness to treatment
Sleep Condition Indicator (SCI) | baseline - 3 months - 9 months
  SCI - 8 item scale evaluating symptoms of insomnia based on DSM 5 criteria
International Physical Activity Questionnaire short form (IPAQ) | baseline - 3 months - 9 months
  IPAQ - surveillance tool assessing levels of physical activity in patients with schizophrenia
Quality of life (S-QoL) | baseline - 3 months - 9 months
  (S-QoL) - self-assessment questionnaire assessing health related quality of life in schizophrenic populations
Functional Remission of General Schizophrenia (FROGS) | baseline - 3 months - 9 months
  FROGS - 19 item questionnaire assessing level of functional remission in schizophrenic populations
Intrinsic Motivation Inventory for Schizophrenia Research (IMI-SR) | baseline - 3 months - 9 months
  IMI-SR - self-report scale with 21 items evaluating intrinsic motivation in schizophrenic populations
French National Adult Reading Test (fNART) | baseline - 9 months
  fNART - test used in assessing intellectual levels within French speaking populations
California Verbal Learning Test (CVLT) | baseline - 9 months
  CVLT - neuropsychological assessment evaluating episodic verbal learning and memory
Trail Making Test (TMT) | baseline - 9 months
  TMT - neuropsychological assessment evaluating executive functioning (attention, visual exploration, speed, mental flexibility)
Pedometer | baseline - 3 months - 9 months (each time pedometer will be worn during one week)
  Pedometer - electronic portable device - assessment of distance travelled -
Physical examinations (PE) and vital signs (VS) | baseline - 3 months - 9 months
  PE includes - weight, BMI, abdominal perimeter VS includes: heart rate, and arterial blood pressure
Blood samples | baseline - 3 months - 9 months
  lipids, glycaemia, CRP (C-reactive protein)
Microbial translocation | baseline - 3 months - 9 months
  DNA extraction and analyze of LBP (Lipopolysaccharide Binding Protein), CD14s, l'I-FABP (fatty acid-binding proteins), zonulin, real-time PCR (polymerase chain reaction) analysis (DNA16s)
Inflammatory status | baseline - 3 months - 9 months
  GM-CSF (granulocyte-macrophage colony-stimulating factor), IFN-γ, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, TNF-α
Letter-Number Sequencing subtest (LNS) | baseline - 9 months
  good predictor of fluid intelligence and strongly correlates with laboratory working memory measures.

OTHER OUTCOMES:
Activity agenda | baseline - 3 months - 9 months
  level of activities performed will be monitored through weekly agendas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Raffard S, Rainteau N, Bayard S, Laraki Y, Norton J, Capdevielle D. Assessment of the efficacy of a fatigue management therapy in schizophrenia: study protocol for a randomized, controlled multi-centered study (ENERGY). Trials. 2020 Sep 17;21(1):797. doi: 10.1186/s13063-020-04606-6. PMID 32943079